CLINICAL TRIAL: NCT03454269
Title: Role of Retina in Mechanisms of Illusions and Visual Hallucinations Observed in Idiopathic Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-380; 2017-A02605-18 (Other: 2017-A02605-18)
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Parkinson's Disease; Visual Hallucinations
Keywords: Parkinson disease; Visual Hallucinations; Illusions; Retina
MeSH Terms: conditions — Parkinson Disease; Hallucinations; Illusions | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD patients with visual hallucinations (PD-VH) (Active Comparator): PD patients without hallucinations or illusions
  Interventions: Diagnostic Test: Optical Coherence Tomography
- Patients with illusions (PD-I) (Active Comparator): PD patients with Illusions and without hallucinations
  Interventions: Diagnostic Test: Optical Coherence Tomography
- Patients without visual hallucinations or illusions (PD-nVHI)) (Active Comparator): PD patients without Illusions and with hallucinations
  Interventions: Diagnostic Test: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — The Optical Coherence Tomography is a painless analysis without contact with the eye. Patients are sitting in front of the machine. Each eye is analyzed. By a laser scanning system, longitudinal sections of the retina are made at the level of the macula and the optic nerve. The device automatically segments the different layers which are then measurable (in microns) by the ophthalmologist (duration of the analysis: 3 minutes).

SUMMARY:
Parkinson's disease is characterized not only by motor symptoms but also by psycho-behavioral symptoms including Visual Hallucinations (VH) and illusions (I), that are generally associated with a severe functional impairment and a bad prognosis for patients. Visual Hallucinations are defined by a visual perception without any real objet to perceive, whereas illusions are defined by a wrong perceptions of an object that is really present. In most of studies investigating the pathophysiology of VH in PD, no difference is made between VH and I, however different mechanisms could lead to the emergence of these two phenomenon, with different prognosis.

Investigator hypothesize that illusions could be related to a visual impairment, maybe at the retinal level, known to be impaired in PD, whereas Visual hallucinations would be due to a more widespread impairment affecting higher levels visuo-perceptive and cognitive functions.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disorder characterized by tremor, rigidity and akinesia, but patients can also present various non-motor symptoms in the course of their illness, including visual hallucinations, delusions or illusions. Visual Hallucinations are false perceptions (no external stimulus is present; generally caused by internal stimulations), whereas illusions are defined by a wrong perception (an external stimulus is always present). Delusions are false believes .The occurrence of hallucinations in PD is of major importance as it has been shown to be associated with an increased risk of cognitive impairment and could lead to nursing home placement and to increased mortality. It is generally believed that delusions/illusions also imply a bad prognosis with time . However recent data suggest that delusions/illusion are not associated with such a poor outcome regarding cognitive functions and mortality compared to hallucinations suggesting different pathological mechanisms and anatomical substrates . Also, a recent study analyzing the neuropsychological correlates of minor hallucinations in PD did not find executive dysfunction to contribute to the onset of minor psychotic phenomena, but was specifically implicated in the progression to well-structured VH.

Thus illusions and minorVH may have a different pathogenesis and a different prognosis compared to complex VH, however studies exploring the structural and functional changes associated with hallucinations in PD have mainly included patients with well-structured VH and moderate to severe cognitive impairment , making it difficult to define early abnormalities associated with minor hallucinations or illusions.

Several hypotheses are proposed regarding the emergence of hallucinations in PD.

* It has been first suggested that hallucinations in PD could be mainly the result of a chronic exposition to dopaminergic therapy . However, the description of hallucination in untreated PD patients goes against that solely explication . Besides, no strong link has been identified between the occurrence of VH and the dosage and duration of dopaminergic treatment . This suggests that Dopaminergic treatment would not directly cause VH but could be a precipiting factor.
* Sleep-wake cycle disturbances have also been reported as risk factors for the occurrence of VH in PD , and particularly the presence of REM Sleep behavior disorders (RBD) . The emergence of VH in PD patients coinciding with daytime episodes of REM sleep may be dream imagery occurring during wake , however this hypothesis is still debated.
* Other risk factors have been associated with VH in PD such as the disease duration, motor symptom severity and mostly cognitive impairment. Indeed, VH occur mainly in PD patients with cognitive decline , but also VH are predictive of dementia . In fact, cognitive impairment in PD patients, and particularly visuoperceptive impairment, would lead to an impaired processing of visual information. Indeed, impaired frontal and parietal cortical activation have been reported in PD patients with VH while being presented visual stimulations, suggesting a diminished answer to external perceptions in posterior cortical areas associated with an increased frontal abnormal activity leading to the emergence of sensorial visual experiences . This shifting visual circuitry from posterior to anterior regions associated with attention process impairment may play a role in the pathophysiology of VH in PD. Thus, the occurrence of Visual Hallucinations in PD Patients appears to be due to a desinhibition of the "top-down" visual stream leading to the emergence of internal mental imagery stocked in memory, and interpreted like visual perceptions coming from the external environment .
* Yet, some evidences also points out to an impaired "bottom-up" processing that could lead to the emergence of VH in PD. Indeed, a dopaminergic denervation and alpha synuclein aggregation have been demonstrated in the retina of PD Patients , even at early stages of the disease . However the functional consequences of such a denervation are still poorly understood , even if impaired contrast discrimination and color vision impairment are widely described in PD . One study has reported an association between retinal impairment, measured with OCT, and VH in PD .

Thus, the emergence of VH and illusions in PD could be due to an inbalance between a hypoactivated "bottom-up" (due to retino-striato-occipital hypoactivation) and a deshinibited "top-down" (mainly frontal) visual stream. However in all these studies, Hallucinations and illusions were not specifically discriminated and investigated in spite of the fact that they could be subtended by different pathophysiological mechanisms and might imply different prognosis for the evolution of the disease.

Investigator hypothesize that illusions, which represent the failure to successfully integrate stimuli that have been physically presented, could be more related to "bottom up" impairment, unlike Hallucinations, which occur where there is perception in the absence of any stimulus and could be more related to a "top down" impairment. Thus, PD patients with illusions (PD-I) might present greater retinal degeneration measured by OCT compared to PD patients with Visual hallucinations (PD-VH) and PD patients without Hallucinations or illusion (PD-nVHI), suggesting a sensorial deprivation underlying these disturbed visual perceptions of reality. Visual Hallucinations that are more elaborated would require a more widespread cognitive disorder, with increased cognitive and visuoperceptive dysfunction.

OBJECTIVE In this study investigator aim to compare PD patients with visual hallucinations (PD-VH), with illusions (PD-I), without Visual hallucinations or illusions (PD-nVHI) regarding retinal degeneration in OCT and cognitive functions (visuoperceptive and attentional functions) in order to determine whether PD-I might show greater retinal degeneration compared to PD-VH, and lesser cognitive impairment.

DESIGN OF STUDY:

Investigator will include 30 PD-VH+, 30 PD-I+, 30 PD-VH-I- among the patients consulting at our center.

During the first visit (Baseline, inclusion visit, 2 hours), each subject will perform a clinical and neurological examination with : • Diagnosis of PD according to UKPDBB criteria.

• The presence of Visual Hallucinations or Illusions will be characterized according to the Psychosensory Hallucination Scale. Illusions will be defined by answering "Yes" to at least one of the "elementary items".

During the second visit (Day 15, one day), each patient will have a neurological, neuropsychological and ophthalmological examination with an evaluation of

* the severity of the disease (Hoehn and Yahr score, Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS))
* the cognitive impairment (Montreal Cognitive Assessment, Evaluation of visuo-perceptive functions and attention)
* the excessive diurnal Somnolence and sleep attacks
* the visual acuity, intraocular pressure, Optical Coherence Tomography (OCT), contrast and colour evaluations.

Circumstances of emergence and distress caused by Hallucinations/illusions was also evaluated by measurement of heart rate variability, electrodermal recording, spy glasses and self-evaluation of Stress.

Finally, each subject will have a Magnetic Resonance Imaging (MRI) acquisition.

ELIGIBILITY:
Inclusion Criteria:

* - patients presenting with a Parkinson's Disease according to UKPDSBB criteria
* Patients affiliated to a health insurance company.
* HV-/IV+ Group : patients presenting illusions criteria according to SCOPA, with no visual hallucinations
* HV+/IV- Group : patients presenting visual hallucinations (SCOPA) without illusions
* HV-/IV- Group : patients without hallucinations or illusions SCOPA)

Exclusion Criteria:

* Patients with other neurological diseases than PD.
* Patients with active psychiatric pathologies (psychosis).
* Patients unable to remain sit and still during different ophtalmological exams due to camptocormia and dyskinesias.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Total and segmental Retinal thickness (in microns) measured with Optical Coherence Tomography | at day 15
  Measurement of different retinal layers using Optical coherence tomography

SECONDARY OUTCOMES:
Characteristics and severity of hallucinations/illusions using Psychosensory Hallucination Scale | at baseline
  Four domains (auditory, visual, olfactory and gustatory, cenesthetic hallucination modalities) are defined with nonoverlapping items
Characteristics and severity of hallucinations/illusions measured using the University of Miami Parkinson's Disease Hallucinations Questionnaire | at baseline
Cognitive function evaluated by the Montreal Cognitive Assessment | at day 15
Dementia evaluated by the Mattis Dementia Rating Scale | at day 15
  It generates five subscale scores in the areas of Attention, Initiation-Perseveration, Construction, Conceptualization, and Memory.
Best corrected visual acuity measured by Parinaud scale | at day 15
  Parinaud scale measures the best corrected near visual acuity, the best outcome is P2 and the worth <P24.
Intraocular pressure measured with air pulse tonometer | at day 15
Contrast sensitivity measured using the Vistech test | at day 15
Color vision measured using the Test 15 Hue de Farnsworth | at day 15
Parkinsonian syndrome severity measured with the MDS UPDRS Scale | at day 15
  The full MDS-UPDRS contains questions/evaluations, divided across Part I (Non-Motor Aspects of Experiences of Daily Living), Part II (Motor Aspects of Experiences of Daily Living), Part III (Motor Examination : 33 scores based on 18 items, several with right, left or other body distribution scores), and Part IV (Motor Complications).
Parkinsonian syndrome severity measured by the Hoehn and Yahr score | at day 15
Sleep quality measured by the Parkinson's Disease Sleep Scale | at day 15
  This scale allows to self-rate and quantify the level of sleep disruption being experienced. It rates 15 items that have 0 to 4 options, 4 is the worth option.
Vigilance measurement and sleep Attack research using the Epworth test | at day 15
Volume of grey matter area (frontal , parietal, occipital, mesencephalic cortex area ) measured at the time of Magnetic Resonance Imaging | at day 15
Emergence of Hallucinations/illusions and distress measured by heart rate variability | at day 15
Emergence of Hallucinations/illusions and distress measured by electro dermal recording | at day 15
Emergence of Hallucinations/illusions and distress measured by self-evaluation of Stress questionnaire | at day 15
Emergence of Hallucinations/illusions and distress measured by spy glasses questionnaire | at day 15

CONTACTS AND LOCATIONS:
Overall Officials: Ana MARQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Marques A, Beze S, Lambert C, Bonamy L, de Chazeron I, Rieu I, Chiambaretta F, Durif F. Psycho-sensory modalities of visual hallucinations and illusions in Parkinson's disease. Rev Neurol (Paris). 2021 Dec;177(10):1228-1236. doi: 10.1016/j.neurol.2021.04.007. Epub 2021 Jul 5. PMID 34238577